CLINICAL TRIAL: NCT03806985
Title: Safety and Efficacy of Psilocybin for the Treatment of Headache Disorders: Sub-Study II
Brief Title: Effects of Psilocybin in Concussion Headache
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Challenging to recruit qualifying subjects
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1607018057.B
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Post-Traumatic Headache
Keywords: psilocybin
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo/Low Dose Psilocybin (Experimental): Subjects in this arm receive placebo in the first session and low dose psilocybin in the second session.
  Interventions: Drug: Placebo oral capsule; Drug: Low Dose Psilocybin
- Placebo/High Dose Psilocybin (Experimental): Subjects in this arm receive placebo in the first session and high dose psilocybin in the second session.
  Interventions: Drug: Placebo oral capsule; Drug: High Dose Psilocybin
- Low Dose Psilocybin/Placebo (Experimental): Subjects in this arm receive low dose psilocybin in the first session and placebo in the second session.
  Interventions: Drug: Placebo oral capsule; Drug: Low Dose Psilocybin
- High Dose Psilocybin/Placebo (Experimental): Subjects in this arm receive high dose psilocybin in the first session and placebo in the second session.
  Interventions: Drug: Placebo oral capsule; Drug: High Dose Psilocybin
- High Dose Psilocybin/Low Dose Psilocybin (Experimental): Subjects in this arm receive high dose psilocybin in the first session and low dose psilocybin in the second session.
  Interventions: Drug: Low Dose Psilocybin; Drug: High Dose Psilocybin
- Low Dose Psilocybin/High Dose Psilocybin (Experimental): Subjects in this arm receive low dose psilocybin in the first session and high dose psilocybin in the second session.
  Interventions: Drug: Low Dose Psilocybin; Drug: High Dose Psilocybin

INTERVENTIONS:
Drug: Placebo oral capsule — microcrystalline cellulose capsule
  Arms: High Dose Psilocybin/Placebo; Low Dose Psilocybin/Placebo; Placebo/High Dose Psilocybin; Placebo/Low Dose Psilocybin
Drug: Low Dose Psilocybin — 0.0143 mg/kg psilocybin capsule (weight-based option) or 1 mg psilocybin capsule (fixed-dose option)
  Arms: High Dose Psilocybin/Low Dose Psilocybin; Low Dose Psilocybin/High Dose Psilocybin; Low Dose Psilocybin/Placebo; Placebo/Low Dose Psilocybin
Drug: High Dose Psilocybin — 0.143 mg/kg psilocybin capsule (weight-based option) or 10 mg psilocybin capsule (fixed-dose option)
  Arms: High Dose Psilocybin/Low Dose Psilocybin; High Dose Psilocybin/Placebo; Low Dose Psilocybin/High Dose Psilocybin; Placebo/High Dose Psilocybin

SUMMARY:
The purpose of this study is to investigate the effects of oral psilocybin in post-traumatic headache. Subjects will be randomized to receive placebo, low dose psilocybin, or high dose psilocybin on two separate test days approximately 14 days apart. Subjects will maintain a headache diary prior to, during, and after the treatments in order to document headache frequency and intensity, as well as associated symptoms. Blood samples will be drawn at various timepoints to measure levels of inflammatory peptides.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of post-traumatic headache
* Typical pattern of headache attacks with approximately two attacks or more weekly
* Attacks are managed by means involving no more than twice weekly triptan use

Exclusion Criteria:

* Axis I psychotic disorder (e.g. schizophrenia, bipolar I, depression with psychosis)
* Axis I psychotic disorder in first degree relative
* Unstable medical condition, severe renal, cardiac or hepatic disease, pacemaker, or serious central nervous system pathology
* Pregnant, breastfeeding, lack of adequate birth control
* History of intolerance to psilocybin, LSD, or related compounds
* Drug or alcohol abuse within the past 3 months (excluding tobacco)
* Urine toxicology positive to drugs of abuse
* Use of vasoconstrictive medications (i.e. sumatriptan, pseudoephedrine, midodrine) within 5 half-lives of test days
* Use of serotonergic antiemetics (i.e. ondansetron) in the past 2 weeks
* Use of antidepressant medication (i.e. TCA, MAOI, SSRI) in the past 6 weeks
* Use of steroids or certain other immunomodulatory agents (i.e. azathioprine) in the past 2 weeks

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Acute change in pain intensity | Measured at 0, 1, 2, 4, and 24 hours after drug administration
  4-tiered pain score (0=none, 1=mild, 2=moderate, 3=severe)
Acute change in nausea/vomiting | Measured at 0, 1, 2, 4, and 24 hours after drug administration
  4-tiered pain score (0=none, 1=mild, 2=moderate, 3=severe)
Acute change in photophobia | Measured at 0, 1, 2, 4, and 24 hours after drug administration
  4-tiered pain score (0=none, 1=mild, 2=moderate, 3=severe)
Acute change in phonophobia | Measured at 0, 1, 2, 4, and 24 hours after drug administration
  4-tiered pain score (0=none, 1=mild, 2=moderate, 3=severe)
Acute change in functional disability | Measured at 0, 1, 2, 4, and 24 hours after drug administration
  4-tiered pain score (0=none, 1=mild, 2=moderate, 3=severe)
Time to first headache attack | Two weeks following each test session
  Measured in days
Time to last headache attack | Two weeks following each test session
  Measured in days
Change in headache attack frequency | From two weeks before first session to two weeks after second session using a headache diary
  Average number (number per week)
Change in headache attack duration | From two weeks before first session to two weeks after second session using a headache diary
  Average duration (measured in hours)
Change in pain intensity of headache attacks | From two weeks before first session to two weeks after second session using a headache diary
  Average pain intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of nausea/vomiting during headache attacks | From two weeks before first session to two weeks after second session using a headache diary
  Average intensity of nausea/vomiting (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of photophobia during headache attacks | From two weeks before first session to two weeks after second session using a headache diary
  Average intensity of photophobia (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of phonophobia during headache attacks | From two weeks before first session to two weeks after second session using a headache diary
  Average intensity of phonophobia (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of functional disability during headache attacks | From two weeks before first session to two weeks after second session using a headache diary
  Average intensity of functional disability (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)

SECONDARY OUTCOMES:
Use of abortive/rescue medication | From two weeks before first session to two weeks after second session using a headache diary
  number of times per week
Headache attack-free time | From two weeks before first session to two weeks after second session using a headache diary
  Number of 24 hour days (may be non-consecutive)
Quality of life using the Centers for Disease Control (CDC) Health-Related Quality of Life Scale: Healthy Days Symptoms Module | From two weeks before first session to two weeks after second session using a headache diary
  4 questions scored 0 to 30 each; higher numbers indicate worse quality of life.
  (1) pain-related impairment, (2) mood symptoms, (3) anxiety symptoms, and (4) lack of sleep Percent change for each measure as well as total score (range 0 to 120) will be calculated.
Depression using Patient Health Questionnaire 9 (PHQ-9) | From two weeks before first session to two weeks after second session using a headache diary
  9 question self-report questionnaire to assess the presence of depression-related symptoms. Each question is rated on a scale of 0-3 (0 = Not at all; 1 = Several days; 2 = More than half the days; 3 = Nearly every day). Higher scores indicate greater presence of depression-related symptoms.
  Total score is calculated. Total score 5-9 = minimal symptoms; total score 10-14 = Major Depression, mild; total score 15-19 = Major Depression, moderately severe; total score >20 = Major Depression severe.
Suicide risk using the Columbia Suicide Severity Rating Scale (CSSRS) | From two weeks before first session to two weeks after second session using a headache diary
  A 10-category assessment of suicidal ideation and behavior. 5 categories (scored "yes/no") relate to the presence of suicidal ideation. 5 categories (scored "yes/no") relate to the presence of suicidal behavior. A "yes" to any of the suicidal ideation categories indicates the presence of suicidal ideation; a "yes" to any of the suicidal behavior categories indicates the presence of suicidal behavior.
Psychedelic effects using the 5-Dimensional Altered States of Consciousness (5D-ASC) scale | Taken on each test day approximately 6 hours after drug administration
  94 questions scored 0 to 100 each; higher numbers indicate greater psychedelic effects Questions address 5 dimensions: (1) Oceanic boundlessness (score range 0-2700), (2) Dread of Ego Dissolution (score range 0-2100), (3) Visionary Restructuralization (score range 0-1800), (4) Auditory Alterations (score range 0-1600), and (5) Vigilance reduction (score range 0-1200) Score for each dimension as well as total score (range 0 to 9400) will be measured.
Change in blood pressure | Measured during each test session prior to drug administration, every 15 min in the first hour, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each test day (mmHg)
Change in heart rate | Measured during each test session prior to drug administration, every 15 min in the first hour, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each test day (beats per minute)
Change in peripheral oxygenation | Measured during each test session prior to drug administration, every 15 min in the first hour, every 30 min in the second hour, and then hourly for 4 hours or until resolution of psychedelic effects (~6 hours post drug)
  Maximum change from baseline during each test day (SpO2)
Change in peripheral levels of calcitonin gene-related peptide (CGRP) | Measured during each test session prior to drug administration, and at 2 and 4 hours after drug administration
  Change from baseline during each test day (pg/mg protein)
Change in peripheral levels of pituitary adenylate cyclase-activating peptide (PACAP) | Measured during each test session prior to drug administration, and at 2 and 4 hours after drug administration
  Change from baseline during each test day (pg/mg protein)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States